CLINICAL TRIAL: NCT05701358
Title: A Randomized Trial of Physiology-guided vs Angiography-guided Non-culprit Lesion Complete Revascularization Strategies & an Observational Study of Optical Coherence Tomography in Patients With Acute MI & Multivessel Coronary Artery Disease
Brief Title: Physiology-guided vs Angiography-guided Non-culprit Lesion Complete Revascularization for Acute MI & Multivessel Disease
Acronym: COMPLETE-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COMPLETE-2
Record Dates: First submitted 2023-01-17; First posted 2023-01-27 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Acute Myocardial Infarction; Coronary Artery Disease
Keywords: NSTEMI; STEMI; multi-vessel disease; optical coherence tomography; FFR; RFR; percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease; Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physiology-guided Non-Culprit-Lesion (NCL) PCI (Active Comparator): Patients randomized to this group will have their physiology assessment using RFR and/or FFR of all qualifying NCLs that were identified prior to randomization. Other validated non-hyperemic physiology ratios (eg. iFR) may only be used when RFR is not available.
  Interventions: Procedure: Physiology-guided NCL PCI
- Angiography-guided NCL PCI (Other): Patients randomized to this group will undergo routine staged PCI of all qualifying NCLs that were identified prior to randomization.
  Interventions: Procedure: Angiography-guided NCL PCI

INTERVENTIONS:
Procedure: Physiology-guided NCL PCI — For RFR, PCI will be performed as per local practice for all lesions with RFR ≤0.89. For FFR, PCI will be performed as per local practice for all NCLs with FFR ≤0.80.
  Arms: Physiology-guided Non-Culprit-Lesion (NCL) PCI
Procedure: Angiography-guided NCL PCI — PCI will be performed as per local practice
  Arms: Angiography-guided NCL PCI

SUMMARY:
COMPLETE-2 is a prospective, multi-centre, randomized controlled trial comparing a strategy of physiology-guided complete revascularization to angiography-guided complete revascularization in patients with acute ST-segment elevation myocardial infarction (STEMI) or non-ST-segment elevation myocardial infarction (NSTEMI) and multivessel coronary artery disease (CAD) who have undergone successful culprit lesion Percutaneous Coronary Intervention (PCI).

COMPLETE-2 OCT is a large scale, prospective, multi-centre, observational, imaging study of patients with STEMI or NSTEMI and multivessel CAD in a subset of eligible COMPLETE-2 patients.

DETAILED DESCRIPTION:
COMPLETE-2 STUDY OBJECTIVES

1. To determine whether a strategy of physiology-guided complete revascularization is non-inferior to a strategy of angiography-guided complete revascularization on the efficacy composite outcome of cardiovascular (CV) death, new myocardial infarction (MI) or ischemia-driven revascularization (IDR).
2. To determine whether a physiology-guided complete revascularization strategy is superior to an angiography-guided complete revascularization strategy in reducing the safety composite outcome of clinically significant bleeding, stroke, stent thrombosis or contrast-associated acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with STEMI or type 1 NSTEMI and within 72 hours of successful culprit-lesion PCI
2. Residual coronary artery disease defined as at least 1 additional non-infarct-related coronary artery stenosis that meets all of the following criteria:

   1. Amenable to successful treatment with PCI
   2. At least 50% diameter stenosis by visual estimation
   3. At least 2.5 mm in diameter
3. Planned complete revascularization strategy for qualifying MI

Exclusion Criteria:

1. Planned or prior coronary artery bypass graft (CABG) surgery
2. Inability to clearly identify a culprit lesion for STEMI or NSTEMI based on angiographic appearance and/or ECG changes and/or regional wall motion abnormalities
3. Prior PCI of a non-culprit lesion in a different vessel from the culprit lesion within 45 days of randomization
4. Planned medical treatment of all qualifying non-culprit lesions (i.e., no PCI)
5. Presence of severe non-culprit-lesion stenosis with reduced epicardial flow (TIMI flow ≤ 2) or >90% visual diameter stenosis
6. Presence of a chronic total occlusion (CTO) if it is the only qualifying non-culprit lesion (patients with a CTO plus additional qualifying non-culprit lesions are eligible)
7. The only qualifying non-culprit lesion is in the same vessel territory as the culprit lesion
8. Baseline STEMI or NSTEMI was due to a suspected non-atherothrombotic mechanism such as type 2 MI (supply-demand mismatch), including spontaneous coronary artery dissection or coronary artery embolism
9. Non-cardiovascular co-morbidity with expected life expectancy <2 years
10. Any other medical, geographic, or social factor making study participation impractical or precluding 5 year follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5100 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Time to first occurrence of the composite of CV death, new MI, or IDR | at study completion, a minimum of 2 years
Safety: Time to first occurrence of the composite of clinically significant bleeding, stroke, stent thrombosis, or contrast-associated acute kidney injury. | at study completion, a minimum of 2 years

SECONDARY OUTCOMES:
Time to first occurrence of the composite of CV death or new MI. | at study completion, a minimum of 2 years
Net clinical outcome: Time to first occurrence of the composite of CV death, new MI, clinically significant bleeding, stroke, stent thrombosis or contrast-associated acute kidney injury. | at study completion, a minimum of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shamir Mehta, MD, Principal Investigator — Population Health Research Institute
Locations (113):
- United States (13):
  - UCLA, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Cardiovascular Research Institute of Kansas, Wichita, Kansas
  - The Johns Hopkins University School of Medicine, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Metropolitan Cardiology Consultants / Metropolitan Heart and Vascular Institute (MCC/MHVI), Coon Rapids, Minnesota
  - RWJ Barnabas Health, Jersey City, New Jersey
  - Bassett Medical Center, Cooperstown, New York
  - VA New York Harbor HealthCare System, New York, New York
  - NYU Grossman School of Medicine, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Virginia Medical Center, Charlottesville, Virginia
- Westmead Hospital, Westmead, New South Wales, Australia
- Klinik Floridsdorf, Vienna, Austria
- Canada (24):
  - McGill University Health Centre (MUHC), Montreal, Quebec
  - William Osler Health System, Brampton
  - University of Alberta Hospital, Mazankowski Heart, Edmonton
  - Hamilton Health Sciences, Hamilton
  - Kingston Health Sciences Centre, Kingston
  - St. Mary's General Hospital, Kitchener
  - London Health Sciences Centre, London
  - Centre Hospitalier de l'Universite de Montreal, Montreal
  - Hopital du Sacre-Coeur de Montreal, Montreal
  - Southlake Regional Health Centre, Newmarket
  - Nova Scotia Health, Nova Scotia
  - University of Ottawa Heart Institute, Ottawa
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec
  - Regina General Hospital, Regina
  - Royal University Hospital, Saskatoon
  - Niagara Health, St. Catharines
  - Newfoundland and Labrador Health Services, St. John's
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay
  - St. Michael's Hospital (Unity Health Toronto), Toronto
  - Sunnybrook Health Sciences Centre, Toronto
  - Ciusss McQ - Chaur, Trois-Rivières
  - St Paul's Hospital, Vancouver
  - Vancouver General Hospital, Vancouver
  - St. Boniface Hospital, Winnipeg
- St. Anne's University Hospital, Brno, Czechia
- Denmark (3):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet - Copenhagen University Hospital, Copenhagen
- Finland (3):
  - Helsinki University Hospital, Helsinki
  - TAYS Sydankeskus Oy, Tampere
  - Turku University Hospital, Turku
- Germany (7):
  - St. Vinzenz-Hospital, Cologne
  - Helios Amper-Klinikum, Dachau
  - Universitatsklinikum Frankfurt, Frankfurt
  - Marienkrankenhaus, Hamburg
  - Schoen Klink Hamburg, Hamburg
  - University Heart & Vascular Center Hamburg, Hamburg
  - WKK Heide, Heide
- Hungary (2):
  - Gottsegen National Cardiovascular Center, Budapest
  - University of Szeged, Szeged
- India (10):
  - Lisie Hospital, Ernākulam, Kerala
  - Meditrina Hospital, Kollam, Kerala
  - Caritas Hospital Trust, Kottayam, Kerala
  - Apollo Rajshree Hospitals, Indore, Madhya Pradesh
  - Rukmani Birla Hospital, Jaipur, Rajasthan
  - Apollo Hospital, Chennai, Tamil Nadu
  - The Madras Medical Mission, Chennai, Tamil Nadu
  - Meenakshi Mission Hospital and Research Center, Madurai, Tamil Nadu
  - Medicover Hospitals, Hyderabad
  - Krishna Institute of Medical Sciences, Secunderabad
- Italy (6):
  - Azienda USL Toscana Sud Est, Arezzo
  - UOC Cardiologia - Ospedale Maggiore, Bologna
  - Azienda Ospedaliero - Universitaria di Ferrara, Ferrara
  - Misericordia Hospital, Grosseto
  - Azienda USL-IRCCS di Reggio Emilia, Reggio, Reggio Emilia
  - Sant Andrea Hospital - Sapienza University, Rome
- Norway (4):
  - Sorlandet Hospital Arendal, Kristiansand, Arendal
  - Oslo University Hospital Ulleval, Oslo
  - Stavanger University Hospital, Stavanger
  - University Hospital Tromso, Tromsø
- Poland (3):
  - Provincial Specialized Hospital, Legnica, Lower Silesian Voivodeship
  - Miedziowym Centrum Zdrowia S.A. w Lubinie, Lubin, Lower Silesian Voivodeship
  - Medical University of Warsaw, Warsaw, Masovian Voivodeship
- Serbia (2):
  - Institute for Cardiovascular Diseases Dedinje, Belgrade
  - University Clinical Center of Serbia, Belgrade
- Spain (7):
  - Hospital Clinico San Carlos, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Clinico Universitario de Valladolid, Valladolid
- Sweden (7):
  - Karolinska University Hospital, Huddinge
  - Lanssjukhuset RYHOV, Jönköping
  - Karlstad Central Hospital, Karlstad
  - Skane University Hospital, Lund
  - Danderyd Hospital, Stockholm
  - Umeå University Hospital, Umeå
  - Uppsala University Hospital, Uppsala
- United Kingdom (19):
  - East Kent Hospitals University NHS Foundation Trust, Ashford
  - Blackpool Teaching Hospitals, Blackpool
  - Ninewells Hospital, Dundee
  - Harefield Hospital, Harefield
  - Kettering General Hospital, Kettering
  - University Hospitals of Leicester, Leicester
  - Liverpool Heart and Chest Hospital, Liverpool
  - Barts Health NHS Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Royal Free London NHS Foundation Trust, London
  - Manchester University NHS Foundation Trust, Manchester
  - The James Cook University Hospital, Middlesbrough
  - Freeman Hospital, Newcastle upon Tyne
  - Royal Berkshire Foundation NHS Trust, Reading
  - Sheffield Teaching Hospitals, Sheffield
  - East and North Hertfordshire NHS Trust, Stevenage
  - Royal Cornwall Hospitals NHS Trust, Truro
  - The Royal Wolverhampton NHS Trust, Wolverhampton
  - Worcestershire Acute Hospitals NHS Trust, Worcester

IPD SHARING:
Plan to Share IPD: No